CLINICAL TRIAL: NCT02351193
Title: A Predictive Scheme to Assess the Outcome of IVF/ICSI Cycles in Poor Responders. an Observational Study in Egypt
Brief Title: a Predictive Scheme for Poor Responders in IVF Cycles
Status: Completed | Type: Observational
Sponsor: Dina Mohamed Refaat Dakhly (Other)
Responsible Party: Sponsor-Investigator, Dina Mohamed Refaat Dakhly, Lecturer of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Organization: Woman's Health University Hospital, Egypt (Other)
Other Study IDs: 26012015
Record Dates: First submitted 2015-01-26; First posted 2015-01-30 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: poor responder females with age less than 35
  Interventions: Other: transvaginal Ultrasound
- Group II: poor responder females with age more than 35
  Interventions: Other: transvaginal Ultrasound

INTERVENTIONS:
Other: transvaginal Ultrasound

SUMMARY:
While practicing the different assisted reproductive techniques, the investigators are faced daily by the problem of poor responder females, and the debate about predicting its results based on the outcome of the different ORTs used. Due to the cost of AMH as an indicator for ovarian response, the need to re-assess its role was essential in our community, which led us to conduct this prospective multi-center IVF study.

ELIGIBILITY:
Inclusion Criteria:

* normal body mass index (BMI)
* AMH from 0.5-1.1 ng/ml.
* previous history of ≤3 oocytes retrieved using conventional long stimulation protocol

Exclusion Criteria:

* Females suffering from other causes of infertility as tubal, uterine factors or known cases of endometriosis
* severe cases of male factor as azospermia
* females who were unable or not willing to participate in the study were excluded from the study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Poor responder females
Sampling Method: Non-Probability Sample
Enrollment: 928 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of MII oocytes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dina MR Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt